CLINICAL TRIAL: NCT02886741
Title: Evaluation of a Multi-modal Network to Spread an Enhanced SSI Prevention Bundle
Brief Title: A Ten-state Cluster-randomized Controlled Trial of the Institute for Health Improvement's Project JOINTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Institute for Healthcare Improvement (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2010-0488-CR05
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Disorder of Hip Region
Keywords: campaign; surgical site infection; orthopedic surgery; quality improvement; infection control
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quality Improvement Campaign (Other): IHI designed and encouraged implementation of a five-component "enhanced" surgical site infection (SSI) prevention bundle with three relatively new evidence-based practices and two Surgical Care Improvement Program (SCIP) practices.
  The campaign recruited state organizations to share information about evidence-based practices and publicize IHI activities and intervention materials (a "How-to Guide," evidence reviews, a summary of the "business case" for interventions, and tip sheets for surgeons, other providers, patients and families). A project website and email listserv offered learning opportunities including webinar calls, faculty-led office hours, and town hall meetings.
  Interventions: Other: Quality Improvement Campaign
- Comparison (No Intervention): Matched state pairs received no campaign intervention and experienced usual care

INTERVENTIONS:
Other: Quality Improvement Campaign — "How To Guide" addressed development of a QI plan; small-scale tests of change- ("PDSA cycles") to refine implementation approaches through iterative learning; and reliance on multi-disciplinary implementation teams. IHI recruited relevant professional organizations to identify faculty.
  Arms: Quality Improvement Campaign

SUMMARY:
In 2011, IHI designed a new campaign to accelerate uptake of evidence-based practices that had been shown to prevent surgical site infections (SSI) associated with hip and knee arthroplasty. Project JOINTS (Joining Organizations IN Tackling SSIs was a multi-faceted, disciplined initiative that used the Rapid Spread Network (defined above), methods and tools developed during previous IHI campaigns to influence orthopedic practices and hospitals performing hip and knee arthroplasty. Rather than launch nationally as other campaigns have done, Project JOINTS was introduced in a cluster-randomized fashion to enable a rigorous, independent evaluation of its effectiveness in promoting uptake of new evidence-based practices.

DETAILED DESCRIPTION:
For Project JOINTS, the evaluation team designed a state-level cluster randomized trial involving five pairs of states selected and matched on characteristics described below. One state from each pair received the 6-month Project JOINTS campaign, while the other state served as a control. To measure changes in the relevant evidence-based practices, RAND conducted a survey of orthopedic surgical staff in all ten states before and after Project JOINTS. The project was reviewed and approved by the RAND Institutional Review Board.

Intervention: Project JOINTS built on the notion of synergistic use of evidence-based practices.14 IHI designed and encouraged implementation of a five-component "enhanced" SSI prevention bundle included three relatively new evidence-based practices and two well-established Surgical Care Improvement Program (SCIP) practices. The three evidence-based practices not consistently implemented by hospitals prior to 2010 were:

1. Screen patients for nasal Staphylococcus aureus (SA) carriage and decolonize SA carriers with five days of intranasal mupirocin and CHG bathing (minimum 3 consecutive days of daily use) in the days immediately preceding surgery;
2. Instruct patients, regardless of SA carriage, to bathe or shower with chlorhexidine gluconate (CHG) for at least three days before surgery;
3. Use an alcohol-containing antiseptic agent for preoperative skin preparation. The campaign recruited state organizations from the RSN developed during the 100,000 Lives and 5 Million Lives Campaigns. The state organizations reached out to hospitals in their states inviting them to participate in the campaign, disseminating information about the campaign and its evidence-based practices, and assisting IHI in publicizing activities described below and in a prior publication.

IHI developed a logic model summarizing how campaign activities were designed to achieve specified goals and this was discussed and refined in collaboration with the evaluation team in order to inform evaluation measures. IHI developed intervention materials (including a "How-to Guide," evidence reviews, a summary of the "business case" for the interventions to prevent SSIs, and tip sheets for surgeons and other providers, and patients and families), created and maintained a project website and email listserv, and offered a range of learning opportunities (including webinar calls, faculty-led office hours, and town hall meetings). Hospital and practice staff who participated in Project JOINTS (typically quality or safety improvement leaders and staff with oversight of infection prevention) received access to a password-protected IHI website maintained by IHI.

In addition to SSI prevention in hip and knee arthroplasty, the Project JOINTs "How To Guide" also addressed important elements of the "Model for Improvement," developed by Associates in Process Improvement and later adapted by IHI for use in its campaigns. These elements included: (1) the development of a QI plan (including explicit aims and a measurement framework); (2) small-scale tests of change- ("PDSA cycles") to refine implementation approaches through iterative learning; and (3) reliance on multi-disciplinary implementation teams. To enhance credibility with clinicians, IHI collaborated with relevant professional organizations, recruiting faculty from the American Academy of Orthopedic Surgeons (AAOS) and the American Association of Hip and Knee Surgeons (AAHKS) and obtaining endorsement from the AAHKS.

ELIGIBILITY:
Inclusion Criteria:

* Surgeons, nurses, and other staff involved in direct care of patients undergoing hip or knee arthroplasty.
* Staff had to be affiliated with one of 20 hospitals selected at random from among all hospitals in each of 10 states that performed a minimum of 100 hip or knee arthroplasties for Medicare beneficiaries.

Exclusion Criteria:

* Per diem staff

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 549 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Adherence to new evidence based practices | 6 months
  The questions addressed three actions (or subcomponents) constituting the nasal screening and decolonization process (new practice 1): screening for SA (1.a.); mupirocin nasal decolonization for methicillin-resistant SA (MRSA) (1.b.) and mupirocin nasal decolonization for methicillin-sensitive SA (MSSA) (1.c.). It included a question on skin decolonization using CHG (new practice 2) and a question on alcohol-containing antiseptic in the operating room (new practice 3). Respondents were asked to indicate the frequency of use of each practice among patients undergoing hip or knee arthroplasty. Response options ranged from 0 to 100% in 10% increments and a "don't know" option. The survey separated practices one and two, but these may not be effective if not used together.

SECONDARY OUTCOMES:
Adherence to established SCIP practices | 6 months
  The survey also included questions on evidence-based practices previously promoted by an established SSI prevention program (the Surgical Care Improvement Program or SCIP): a question about initiation of perioperative intravenous antibiotics within the appropriate time interval prior to the start of arthroplasty (4.a.), a question about use of intravenous vancomycin for prophylaxis for patients known to be MRSA carriers (4.b.), and a question on use of appropriate hair removal techniques

CONTACTS AND LOCATIONS:
Overall Officials: Eric C Schneider, MD, Principal Investigator — The Commonwealth Fund

IPD SHARING:
Plan to Share IPD: No
Aggregate data provided upon request

REFERENCES:
- [Result] Khodyakov D, Ridgely MS, Huang C, DeBartolo KO, Sorbero ME, Schneider EC. Project JOINTS: what factors affect bundle adoption in a voluntary quality improvement campaign? BMJ Qual Saf. 2015 Jan;24(1):38-47. doi: 10.1136/bmjqs-2014-003169. Epub 2014 Nov 5. PMID 25376449